CLINICAL TRIAL: NCT02114827
Title: Efficacy of a Patient Education Video
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study closed due to slow accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-13-10228; HM20000410 (Other: Office of Research Subject Protection)
Record Dates: First submitted 2014-04-03; First posted 2014-04-15 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Leukemia, Not Otherwise Specified; Malignant Neoplasm
Keywords: Multiple Myeloma
MeSH Terms: conditions — Leukemia; Neoplasms; Multiple Myeloma | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Video (Experimental): Patients will view the 23-minute "Guide to Stem Cell Transplantation" video depicting the HSCT experience
  Interventions: Behavioral: Video
- FAQ Sheet (Active Comparator): Patients will receive HSCT FAQ sheet developed by the NCI at the NIH
  Interventions: Behavioral: FAQ Sheet

INTERVENTIONS:
Behavioral: Video — 23-minute video
  Other Names: Guide to Stem Cell Transplantation
  Arms: Video
Behavioral: FAQ Sheet
  Other Names: HSCT Freuently asked questions sheet developed by NCI at NIH
  Arms: FAQ Sheet

SUMMARY:
Patients in the intervention arm will view the 23-minute video depicting the Hematopoietic stem cell transplantation (HSCT) experience. Patients in the control arm will receive HSCT frequently asked questions (FAQ) sheet developed by the National Cancer Institute (NCI) at the National Institutes of Health (NIH).

DETAILED DESCRIPTION:
The study's overall goals are 1) to improve outcomes; and 2) to increase satisfaction with the physician consultation.

Patients will be randomized to intervention or control and data will be collected at three time points (before treatment, 30 days post-HSCT and 12 months post-HSCT).

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients scheduled for HSCT

Exclusion Criteria:

* Patients who have received HSCT previously
* Patients who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in emergency department visits | Up to 12 months after HSCT
  Data will be collected through review of medical and insurance billing records
Change in number of hospitalizations | Up to 12 months after HSCT
  Data will be collected through review of medical and insurance billing records

SECONDARY OUTCOMES:
Perception of satisfaction with the physician consultation | Up to 12 months after HSCT
  The Physician consultation will be measured by the Patient Satisfaction Communication Questionnaire (PSCQA). Participants are asked to rate their experience with the physician consultation. There are 17 items, 8 positively worded and 9 negatively worded. Each item is rated on a 5 point likert scale with 1 being strongly agree to 5 being strongly disagree. The maximum score on the PSCQ is 85. The measure takes approximately 4 minutes to administer.

CONTACTS AND LOCATIONS:
Overall Officials: Robin K Matsuyama, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States